CLINICAL TRIAL: NCT02612207
Title: Validation of Bilirubin Binding Capacity (BBC) Using AVIV Device
Brief Title: Point-of-Care System for Determination of Bilirubin Capacity in Neonates
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Aviv Biomedical, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB-24465
Record Dates: First submitted 2015-11-05; First posted 2015-11-23 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Jaundice, Neonatal; Hyperbilirubinemia; Bilirubin-Induced Neurological Dysfunction (BIND)
Keywords: Bilirubin Binding Capacity Preterm Neonates and Jaundice
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia; Jaundice

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Bilirubin Binding Capacity by Hematofluorometry Validation — Observation study

SUMMARY:
The aims of this observational bench project are to validate the performance of the miniaturized and modernized hematofluorometer that measures bilirubin capacity into a product and is suitable for operation in various point of care environments w in the management of preterm neonates.

DETAILED DESCRIPTION:
The status of bilirubin binding to albumin (Alb) is central to personalized management of unconjugated newborn hyperbilirubinemia, especially those at risk of bilirubin-induced neurologic dysfunction (BIND) (1). Our objectives were to validate the Aviv Bili-4 Hematofluorometer in the context of its usefulness and ease of use based on ad hoc clinical studies and surveys of end-users. In addition, we continued our efforts to validate the Bili-4 device in order to facilitate Aviv, Inc. in their development of claims of the most appropriate use of bilirubin binding capacity (BBC) information in the management of neonates. Neonatal blood samples were obtained from newborns born at Stanford University's LPCH with gestational ages (GA) ranging from 22-40 wks. Total bilirubin (TB), Alb and apparent serum unbound bilirubin (UB) concentrations were measured or calculated. Ratios of bound bilirubin (BB) to reserve Alb binding capacity for bilirubin (RABC) were also determined. Bilirubin binding capacity (BBC) by hematofluorometry (Hmf) was compared to the calculated BBC (or 8.8 × Alb) using Alb levels as measured by the clinical laboratory. We report the progress of this inquiry at the Stanford University (1).

ELIGIBILITY:
Inclusion Criteria are in vitro testing of blood samples obtained from eligible babies:

* Subjects must meet all of the following inclusion criteria to be considered eligible for study enrollment soon after birth or re-admission (for phototherapy):

  * Parental informed consent
  * Male and female newborns with a GA ≥ 24 wks with a birthweight ≥ 500 g as well as sick or unstable late preterm newborns infants with GA ≥ 35 wks with a birthweight ≥ 2500 g.
  * Enrollment at age less than 14 days and more than 6h

Exclusion Criteria:

* None.

Ages: 6 Hours to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of preterm (≥ 24 wks GA, BW≥500g) as well as sick or unstable late-term newborns (infants ≥ 35 wks GA, BW≥2500g).
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Bilirubin Binding Capacity (BBC) on healthy and at-risk infants for impaired binding capacity by hematofluorometery assay | <14 days of life
  To define normative data (mean, median, range, inter-quartile ranges) among these deemed healthy infants (including those who are at- risk) for increased vulnerability to impaired binding soon after birth

SECONDARY OUTCOMES:
Natural history of BBC and stratification of those at risk of disordered bilirubin binding | <14 days of life
  To delineate the prospective natural history of BBC and stratify those at most or least likely at risk of impaired bilirubin binding

CONTACTS AND LOCATIONS:
Overall Officials: Vinod K Bhutani, MD, Principal Investigator — PI
Locations (2):
- United States (2):
  - Lucile-Packard Children's Hospital at Stanford, Stanford, California
  - AVIV Biomedical, Inc., Lakewood, New Jersey

REFERENCES:
- [Result] Lamola AA, Bhutani VK, Du L, Castillo Cuadrado M, Chen L, Shen Z, Wong RJ, Stevenson DK. Neonatal bilirubin binding capacity discerns risk of neurological dysfunction. Pediatr Res. 2015 Feb;77(2):334-9. doi: 10.1038/pr.2014.191. Epub 2014 Nov 24. PMID 25420178